CLINICAL TRIAL: NCT00419640
Title: Septal Pacing for Atrial Fibrillation Suppression Evaluation
Brief Title: SAFE Study - Septal Pacing for Atrial Fibrillation Suppression Evaluation
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR04032AF
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
Keywords: Sinus node disease; AV node disease
MeSH Terms: conditions — Atrial Fibrillation; Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LAS + DAO ON (Experimental): The right atrial lead is placed in the low atrial septal position and the DAO algorithm is turned ON.
  Interventions: Device: Pacemaker implantation with RA lead in LAS position
- LAS + DAO OFF (Experimental): The right atrial lead is placed in the low atrial septal position and the DAO algorithm is turned OFF.
  Interventions: Device: Pacemaker implantation with RA lead in LAS position
- RAA + DAO ON (Experimental): The right atrial lead is placed in the right atrial appendage position and the DAO algorithm is turned ON.
  Interventions: Device: Pacemaker implantation with RA lead in RAA position
- RAA + DAO OFF (Active Comparator): The right atrial lead is placed in the right atrial appendage position and the DAO algorithm is turned OFF.
  Interventions: Device: Pacemaker implantation with RA lead in RAA position

INTERVENTIONS:
Device: Pacemaker implantation with RA lead in LAS position — Pacemaker implantation with RA lead placed in low atrial septal position
  Other Names: Identity ADx DR device
  Arms: LAS + DAO ON
Device: Pacemaker implantation with RA lead in LAS position — Pacemaker implantation with RA lead placed in low atrial septal position
  Other Names: Identity ADx DR pacemaker
  Arms: LAS + DAO OFF
Device: Pacemaker implantation with RA lead in RAA position — Pacemaker implantation with RA lead placed in right atrial appendage position
  Other Names: Identity ADx DR pacemaker
  Arms: RAA + DAO ON
Device: Pacemaker implantation with RA lead in RAA position — Pacemaker implantation with RA lead placed in right atrial appendage position
  Other Names: Identity ADx DR pacemaker
  Arms: RAA + DAO OFF

SUMMARY:
This is a randomized, parallel, single-blinded multi-center study. The objective is to compare the long term clinical outcomes among the site of atrial pacing and to compare the long term effect of the atrial fibrillation (AF) Suppression algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. Have a history of paroxysmal AF with documented AF episode within the last 6 months; documentation of AF is required. It can be documented by one of the following:

   * Holter documentation and the strip must be at least 30 seconds; OR
   * one page of 12-lead electrocardiogram (ECG); OR
   * transtelephonic recording for more than 15 seconds.
2. Have a conventional indication for a pacemaker due to either sinus or atrioventricular (AV) node diseases.
3. Provide written informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluations.
4. Be at least 18 years old.

Exclusion Criteria:

1. Already implanted with a pacemaker or implantable cardioverter defibrillator (ICD).
2. Are expected to have heart surgery within the next 6 months.
3. Have angina pectoris, New York Heart Association (NYHA) Class III or Class IV.
4. Are expected not to be able to tolerate high rate pacing.
5. Have less than 12 months' life expectancy.
6. Are on the cardiac transplantation list.
7. Are in chronic AF.
8. Have a reversible aetiology of AF (e.g., hyperthyroidism, acute post-cardiac surgery AF, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2005-05; Primary Completion 2012-02 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Persistent AF and chronic AF | 2 years

SECONDARY OUTCOMES:
Device diagnostic data: number of atrial high rate episode, mode switch episode and AF burden | 2 years
Number of cardioversions | 2 years
Safety and efficacy of low septal pacing | 2 years
Echocardiogram (Echo) parameters include left ventricular ejection fraction (LVEF) and diastolic index using Doppler Echo | 2 years
Quality-of-life questionnaire: Short Form-36 (SF-36) | 2 years
Major cardiovascular events: heart failure, stroke, hospitalization, and cardiovascular mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chu-Pak Lau, Prof., Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, The University Hospital of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lau CP, Tachapong N, Wang CC, Wang JF, Abe H, Kong CW, Liew R, Shin DG, Padeletti L, Kim YH, Omar R, Jirarojanakorn K, Kim YN, Chen MC, Sriratanasathavorn C, Munawar M, Kam R, Chen JY, Cho YK, Li YG, Wu SL, Bailleul C, Tse HF; Septal Pacing for Atrial Fibrillation Suppression Evaluation Study Group. Prospective randomized study to assess the efficacy of site and rate of atrial pacing on long-term progression of atrial fibrillation in sick sinus syndrome: Septal Pacing for Atrial Fibrillation Suppression Evaluation (SAFE) Study. Circulation. 2013 Aug 13;128(7):687-93. doi: 10.1161/CIRCULATIONAHA.113.001644. Epub 2013 Jul 18. PMID 23868858